CLINICAL TRIAL: NCT04329104
Title: Safety and Efficacy of VRC-MALMAB0100-00-AB (CIS43LS), a Human Monoclonal Antibody Against Plasmodium Falciparum, in a Dose-Escalation Trial and a Randomized, Double-Blind Trial of Adults in Mali
Brief Title: Safety and Efficacy of CIS43LS Anti-malaria mAb in Mali
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Malaria Research and Training Center, Bamako, Mali (Other); University of Washington (Other); Harvard School of Public Health (HSPH) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: 2020/32/CE/FMOS/FAPH
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Results first posted 2024-05-02 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Plasmodium Falciparum Infection; Malaria
MeSH Terms: conditions — Malaria | interventions — CIS43LS; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Dose-escalation study: Arm 1: 5 mg/kg of CIS43LS (Experimental): Participants receive 5 mg/kg of CIS43LS as one time intravenous infusion on Day 0.
  Interventions: Biological: VRC-MALMAB0100-00-AB (CIS43LS)
- Dose-escalation study: Arm 2: 10 mg/kg of CIS43LS (Experimental): Participants receive 10 mg/kg of CIS43LS as one time intravenous infusion on Day 0.
  Interventions: Biological: VRC-MALMAB0100-00-AB (CIS43LS)
- Dose-escalation study: Arm 3: 40 mg/kg of CIS43LS (Experimental): Participants receive 40 mg/kg of CIS43LS as one time intravenous infusion on Day 0.
  Interventions: Biological: VRC-MALMAB0100-00-AB (CIS43LS)
- Efficacy study: Arm 1: 10 mg/kg of CIS43LS (Experimental): Participants receive 10 mg/kg of CIS43LS as one time intravenous infusion on Day 0.
  Interventions: Biological: VRC-MALMAB0100-00-AB (CIS43LS)
- Efficacy study: Arm 2: 40 mg/kg of CIS43LS (Experimental): Participants receive 40 mg/kg of CIS43LS as one time intravenous infusion on Day 0.
  Interventions: Biological: VRC-MALMAB0100-00-AB (CIS43LS)
- Efficacy study: Arm 3: Placebo (Placebo Comparator): Participants receive placebo as one time intravenous infusion on Day 0.
  Interventions: Other: Normal saline

INTERVENTIONS:
Biological: VRC-MALMAB0100-00-AB (CIS43LS) — Administered via one-time intravenous infusion
  Arms: Dose-escalation study: Arm 1: 5 mg/kg of CIS43LS; Dose-escalation study: Arm 2: 10 mg/kg of CIS43LS; Dose-escalation study: Arm 3: 40 mg/kg of CIS43LS; Efficacy study: Arm 1: 10 mg/kg of CIS43LS; Efficacy study: Arm 2: 40 mg/kg of CIS43LS
Other: Normal saline — Administered via one-time intravenous infusion
  Arms: Efficacy study: Arm 3: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and efficacy of VRC MALMAB0100-00-AB (CIS43LS), a human monoclonal antibody, against naturally occurring Plasmodium falciparum (Pf) infection.

DETAILED DESCRIPTION:
This study will evaluate the safety, tolerability, and efficacy of VRC MALMAB0100-00-AB (CIS43LS), a human monoclonal antibody, against naturally occurring Plasmodium falciparum (Pf) infection.

The first part of the study is an open-label dose-escalation study for safety and tolerability. Participants will be assigned to one of three dose arms. Dosing will begin in the lowest dose arm. Once all participants in that arm reach Day 7 post-infusion, if no safety concerns have arisen, dosing will begin at the subsequent dose level. This process will be repeated until participants complete the third dose arm. Participants will be followed for safety to assess adverse events (AEs) at study visits 1, 3, 7, 14, 21, and 28 days after administration, then monthly through 24 weeks after administration.

After the last subject in the highest dose arm reaches Day 7 safety follow-up, an interim safety evaluation will be performed before enrollment begins for the second part of the study.

The second part of the study is a randomized, double-blind, placebo-controlled trial to assess safety and protective efficacy of CIS43LS and placebo. Participants in the efficacy study will receive the study agent and be followed at study visits 1, 3, 7, 14, 21, and 28 days later, and once every 2 weeks thereafter through 24 weeks. Primary study assessments include physical examinations and blood collection for identification of Pf infection and other research laboratory evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 and ≤55 years.
* Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
* In good general health and without clinically significant medical history.
* Able to provide informed consent.
* Willing to have blood samples and data stored for future research.
* Resides in or near Kalifabougou or Torodo, Mali, and available for the duration of the study.
* Females of childbearing potential must be willing to use reliable contraception from 21 days prior to study day 0 through the final study visit as described below.

  * Reliable methods of birth control include 1 of the following: confirmed pharmacologic contraceptives via parenteral delivery or intrauterine or implantable device.
  * Nonchildbearing women will be required to report date of last menstrual period, history of surgical sterility (i.e., tubal ligation, hysterectomy) or premature ovarian insufficiency, and will have urine or serum pregnancy test performed per protocol.

Exclusion Criteria:

* Pregnancy, as determined by a positive urine or serum beta-human choriogonadotropin (β-hCG) test (if female).
* Currently breastfeeding.
* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the subject to understand and comply with the study protocol.
* Study comprehension examination score of <80% correct or per investigator discretion.
* Hemoglobin, white blood cell, absolute neutrophil, or platelet count outside the local laboratory-defined limits of normal. (Subjects may be included at the investigator's discretion for "not clinically significant" values.)
* Alanine transaminase (ALT) or creatinine (Cr) level above the local laboratory-defined upper limit of normal. (Subjects may be included at the investigator's discretion for "not clinically significant" values.)
* Infected with human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBV).
* Known or documented sickle cell disease by history. (Note: Known sickle cell trait is NOT exclusionary.)
* Clinically significant abnormal electrocardiogram (ECG; corrected QT interval [QTc] >460 or other significant abnormal findings, including unexplained tachycardia or bradycardia).
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, endocrine, rheumatologic, autoimmune, hematological, oncologic, or renal disease by history, physical examination, and/or laboratory studies including urinalysis.
* Receipt of any investigational product within the past 30 days.
* Participation or planned participation in an interventional trial with an investigational product until the last required protocol visit. (Note: Past, current, or planned participation in observational studies is NOT exclusionary.)
* Medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
* History of a severe allergic reaction or anaphylaxis.
* Severe asthma (defined as asthma that is unstable or required emergent care, urgent care, hospitalization, or intubation during the past 2 years, or that has required the use of oral or parenteral corticosteroids at any time during the past 2 years).
* Pre-existing autoimmune or antibody-mediated diseases including but not limited to: systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjögren's syndrome, or autoimmune thrombocytopenia.
* Known immunodeficiency syndrome.
* Known asplenia or functional asplenia.
* Use of chronic (≥14 days) oral or IV corticosteroids (excluding topical or nasal) at immunosuppressive doses (i.e., prednisone >10 mg/day) or immunosuppressive drugs within 30 days of day 0.
* Receipt of a live vaccine within the past 4 weeks or a killed vaccine within the past 2 weeks prior to study agent administration.
* Receipt of immunoglobulins and/or blood products within the past 6 months.
* Previous receipt of an investigational malaria vaccine in the last 5 years.
* Known allergies or contraindication against artemether-lumefantrine.
* Other condition(s) that, in the opinion of the investigator, would jeopardize the safety or rights of a subject participating in the trial, interfere with the evaluation of the study objectives, or render the subject unable to comply with the protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 348 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2023-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kassoum Kayentao, MD, MPH, PhD, Principal Investigator — Faculté de Médecine Pharmacie d'Odontostomatologie (FMPOS); Peter D. Crompton, MD, MPH, Principal Investigator — National Institutes of Health (NIH)
Locations (2):
- Mali (2):
  - Kalifabougou MRTC Clinic, Kalifabougou, Koulikoro
  - Torodo MRTC Clinic, Torodo, Koulikoro

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kayentao K, Ongoiba A, Preston AC, Healy SA, Doumbo S, Doumtabe D, Traore A, Traore H, Djiguiba A, Li S, Peterson ME, Telscher S, Idris AH, Kisalu NK, Carlton K, Serebryannyy L, Narpala S, McDermott AB, Gaudinski M, Traore S, Cisse H, Keita M, Skinner J, Hu Z, Zeguime A, Ouattara A, Doucoure M, Dolo A, Djimde A, Traore B, Seder RA, Crompton PD; Mali Malaria mAb Trial Team. Safety and Efficacy of a Monoclonal Antibody against Malaria in Mali. N Engl J Med. 2022 Nov 17;387(20):1833-1842. doi: 10.1056/NEJMoa2206966. Epub 2022 Oct 31. PMID 36317783
- [Derived] Skinner J, Kayentao K, Ongoiba A, Healy SA, Hu Z, Preston AC, Niangaly A, Schwabl P, Cisse H, Doumbo S, Doumtabe D, Traore A, Li S, Peterson ME, Seilie AM, Chavtur C, Staubus W, Chang M, Kelley K, Traore H, Djiguiba A, Keita M, Ouattara A, Doucoure M, Keita M, Diarra D, Sylla M, Diakite D, Konate M, Traore S, Zeguime A, Dolo A, Neafsey DE, Murphy SC, Traore B, Seder RA, Crompton PD. Anti-sporozoite monoclonal antibody for malaria prevention: secondary efficacy outcome of a phase 2 randomized trial. Nat Med. 2025 Aug;31(8):2682-2690. doi: 10.1038/s41591-025-03739-y. Epub 2025 Jun 3. PMID 40461818

RESULTS

PARTICIPANT FLOW:
Period: Dose Escalation Study - 5 mg/kg
Arm/Group | Dose-escalation Study: Arm 1: 5 mg/kg of CIS43LS | Dose-escalation Study: Arm 2: 10 mg/kg of CIS43LS | Dose-escalation Study: Arm 3: 40 mg/kg of CIS43LS | Efficacy Study: Arm 1: 10 mg/kg of CIS43LS | Efficacy Study: Arm 2: 40 mg/kg of CIS43LS | Efficacy Study: Arm 3: Placebo
Started | 6 | 0 | 0 | 0 | 0 | 0
Completed | 6 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Dose Escalation Study - 10 mg/kg
Arm/Group | Dose-escalation Study: Arm 1: 5 mg/kg of CIS43LS | Dose-escalation Study: Arm 2: 10 mg/kg of CIS43LS | Dose-escalation Study: Arm 3: 40 mg/kg of CIS43LS | Efficacy Study: Arm 1: 10 mg/kg of CIS43LS | Efficacy Study: Arm 2: 40 mg/kg of CIS43LS | Efficacy Study: Arm 3: Placebo
Started | 0 | 6 | 0 | 0 | 0 | 0
Completed | 0 | 6 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Dose Escalation Study - 40 mg/kg
Arm/Group | Dose-escalation Study: Arm 1: 5 mg/kg of CIS43LS | Dose-escalation Study: Arm 2: 10 mg/kg of CIS43LS | Dose-escalation Study: Arm 3: 40 mg/kg of CIS43LS | Efficacy Study: Arm 1: 10 mg/kg of CIS43LS | Efficacy Study: Arm 2: 40 mg/kg of CIS43LS | Efficacy Study: Arm 3: Placebo
Started | 0 | 0 | 6 | 0 | 0 | 0
Completed | 0 | 0 | 6 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Efficacy Study
Arm/Group | Dose-escalation Study: Arm 1: 5 mg/kg of CIS43LS | Dose-escalation Study: Arm 2: 10 mg/kg of CIS43LS | Dose-escalation Study: Arm 3: 40 mg/kg of CIS43LS | Efficacy Study: Arm 1: 10 mg/kg of CIS43LS | Efficacy Study: Arm 2: 40 mg/kg of CIS43LS | Efficacy Study: Arm 3: Placebo
Started | 0 | 0 | 0 | 110 | 110 | 110
Completed | 0 | 0 | 0 | 105 | 104 | 102
Not Completed | 0 | 0 | 0 | 5 | 6 | 8
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 5 | 6 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose-escalation Study: Arm 1: 5 mg/kg of CIS43LS | Dose-escalation Study: Arm 2: 10 mg/kg of CIS43LS | Dose-escalation Study: Arm 3: 40 mg/kg of CIS43LS | Efficacy Study: Arm 1: 10 mg/kg of CIS43LS | Efficacy Study: Arm 2: 40 mg/kg of CIS43LS | Efficacy Study: Arm 3: Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 110 | 110 | 110 | 348
Age, Customized [Count of Participants; unit: Participants]
  18-20 years | 0 | 1 | 1 | 9 | 13 | 10 | 34
  21-30 years | 1 | 1 | 1 | 34 | 25 | 31 | 93
  31-40 years | 2 | 0 | 1 | 39 | 36 | 41 | 119
  41-50 years | 3 | 4 | 3 | 23 | 34 | 26 | 93
  51-55 years | 0 | 0 | 0 | 5 | 2 | 2 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 51 | 47 | 44 | 149
  Male | 3 | 4 | 4 | 59 | 63 | 66 | 199
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African | 6 | 6 | 6 | 110 | 110 | 110 | 348
Region of Enrollment [Count of Participants; unit: Participants]
  Mali | 6 | 6 | 6 | 110 | 110 | 110 | 348

OUTCOME MEASURES:

1. Primary Outcome: Participants With Local Adverse Events (AEs)
Description: Participants with incidence of local adverse events occurring within 7 days after administration of CIS43LS. Local reactogenicity included pain/tenderness, swelling, redness, bruising, and pruritus at the site of infusion.
Time Frame: Within 7 days after administration of CIS43LS
Population: The analysis included all participants in the dose escalation study.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalation Study: Arm 1: 5 mg/kg of CIS43LS | Dose-escalation Study: Arm 2: 10 mg/kg of CIS43LS | Dose-escalation Study: Arm 3: 40 mg/kg of CIS43LS
Number analyzed (Participants) | 6 | 6 | 6
Participants
  Injection site swelling | 1 | 0 | 0
  Pain at injection site | 2 | 2 | 0
  Tenderness at injection site | 0 | 0 | 0
  Redness at injection site | 0 | 0 | 0
  Bruising at injection site | 1 | 0 | 0
  Pruritus at injection site | 0 | 0 | 0

2. Primary Outcome: Severity of Local Adverse Events (AEs)
Description: The severity of local AEs was graded using the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Clinical Trials.
  Grade 1: Pain = does not interfere with activity; Tenderness = mild discomfort to touch; Erythema/Redness = 2.5-5 cm; Induration/Swelling = 2.5-5 cm and does not interfere with activity.
  Grade 2: Pain = Repeated use of non-narcotic pain reliever > 24 hours or interferes with daily activity; Tenderness = Discomfort with movement; Erythema/Redness = 5.1-10 cm; Induration/Swelling = 5.1-10 cm and interferes with activity.
  Grade 3: Pain = Any use of narcotic pain reliever or prevents daily activity; Tenderness = Significant discomfort at rest; Erythema/Redness = > 10 cm; Induration/Swelling = > 10 cm or prevents daily activity.
  Grade 4: Pain = Emergency room (ER) visit or hospitalization; Tenderness = ER visit or hospitalization; Erythema/Redness = Necrosis or exfoliative dermatitis; Induration/Swelling = Necrosis
  Grade 5: Death
Time Frame: Within 7 days after the administration of CIS43LS
Population: The analysis included all participants in the dose escalation study.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalation Study: Arm 1: 5 mg/kg of CIS43LS | Dose-escalation Study: Arm 2: 10 mg/kg of CIS43LS | Dose-escalation Study: Arm 3: 40 mg/kg of CIS43LS
Number analyzed (Participants) | 6 | 6 | 6
Participants
  Grade 1 | 4 | 2 | 0
  Grade 2 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0

3. Primary Outcome: Participants With Systemic Adverse Events (AEs)
Description: Participants with incidence of systemic adverse events occurring within 7 days after product administration of CIS43LS. Systemic reactogenicity events included fever, feeling unusually tired or unwell, muscle aches, headache, chills, nausea, and joint pain.
Time Frame: Within 7 days after the administration of CIS43LS
Population: The analysis included all participants in the dose escalation study.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalation Study: Arm 1: 5 mg/kg of CIS43LS | Dose-escalation Study: Arm 2: 10 mg/kg of CIS43LS | Dose-escalation Study: Arm 3: 40 mg/kg of CIS43LS
Number analyzed (Participants) | 6 | 6 | 6
Participants
  Fever | 0 | 0 | 0
  Feeling unusually tired or unwell | 0 | 0 | 0
  Muscle aches | 0 | 0 | 0
  Headache | 1 | 1 | 0
  Chills | 0 | 0 | 0
  Nausea | 0 | 0 | 0
  Joint pain | 0 | 0 | 0

4. Primary Outcome: Severity of Systemic Adverse Events (AEs)
Description: The severity of systemic AEs occurring after the administration of CIS43LS was assessed using the grading scale below:
  Grade 1: Fever = 37.5^oC-37.9^oC; Fatigue, Headache, Myalgia = No interference with activity; Nausea = no interference with activity or 1-2 episodes/hour
  Grade 2: Fever = 38^oC-38.4^oC; Fatigue, Myalgia = Some interference with activity; Headache = Repeated use of non-narcotic pain reliever > 24 hours or some interference with activity; Nausea = Some interference with activity or > 2 episodes/24 hours
  Grade 3: Fever = 38.5^oC-39.5^oC; Fatigue = Prevents daily activity; Headache =Significant; any use of narcotic pain reliever or prevents daily activity; Myalgia =Significant; prevents daily activity; Nausea = Prevents daily activity, requires outpatient intravenous hydration
  Grade 4: Fever = > 39.5^oC; Fatigue, Headache, Myalgia = Emergency room (ER) visit or hospitalization; Nausea = ER visit or hospitalization for hypotensive shock
  Grade 5: Death
Time Frame: Within 7 days after the administration of CIS43LS
Population: The analysis included all participants in the dose escalation study.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalation Study: Arm 1: 5 mg/kg of CIS43LS | Dose-escalation Study: Arm 2: 10 mg/kg of CIS43LS | Dose-escalation Study: Arm 3: 40 mg/kg of CIS43LS
Number analyzed (Participants) | 6 | 6 | 6
Participants
  Grade 1 | 1 | 1 | 0
  Grade 2 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0

5. Primary Outcome: Participants With Plasmodium Falciparum (Pf) Infection Detected by Microscopic Examination
Description: Number of participants with Plasmodium falciparum (Pf) blood stage infection defined as blood smear-positive for Pf was assessed by microscopic examination of thick blood smear collected from participants from day 7 through week 24 (168 days) after administration of CIS43LS or placebo. Sample was collected every two weeks until week 24.
Time Frame: Day 7 through week 24 (168 days) after administration of intervention
Population: The analysis included all participants in the efficacy study.
Measure: Count of Participants; unit: Participants
Arm/Group | Efficacy Study: Arm 1: 10 mg/kg of CIS43LS | Efficacy Study: Arm 2: 40 mg/kg of CIS43LS | Efficacy Study: Arm 3: Placebo
Number analyzed (Participants) | 110 | 110 | 110
Participants | 39 | 20 | 86

6. Secondary Outcome: Participants With Plasmodium Falciparum (Pf) Infection Detected by Reverse Transcription Polymerase Chain Reaction (RT-PCR)
Description: Number of participants with Plasmodium falciparum (Pf) blood stage infection defined as blood smear-positive for Pf was assessed by reverse transcription polymerase chain reaction (RT-PCR) using dried blood spot specimen collected from participants from day 21 through week 24 (168 days) after administration of CIS43LS or placebo. Sample was collected every two weeks until 24 weeks. Plasmodium 18S rRNA RT-PCR assay was applied to dried blood spots during analysis.
Time Frame: Day 21 through week 24 (168 days) after administration of intervention
Population: The analysis included all participants in the efficacy study.
Measure: Count of Participants; unit: Participants
Arm/Group | Efficacy Study: Arm 1: 10 mg/kg of CIS43LS | Efficacy Study: Arm 2: 40 mg/kg of CIS43LS | Efficacy Study: Arm 3: Placebo
Number analyzed (Participants) | 110 | 110 | 110
Participants | 48 | 29 | 96

7. Secondary Outcome: Maximum Serum Concentration (Cmax) for CIS43LS
Description: Maximum serum concentration (Cmax) of CIS43LS by dose group following a single intravenous administration to assess durability of CIS43LS and allow for correlation with Plasmodium falciparum (Pf) infection risk. Cmax is the peak serum concentration that CIS43LS achieves after it has been administered. It is determined as a maximum value on the summary pharmacokinetic (PK) curve for each study group and measured by a Meso Scale Discovery LLC-based automation platform.
Time Frame: Measured through Week 24
Population: All participants who received CIS43LS, excluding placebo group.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Dose-escalation Study: Arm 1: 5 mg/kg of CIS43LS | Dose-escalation Study: Arm 2: 10 mg/kg of CIS43LS | Dose-escalation Study: Arm 3: 40 mg/kg of CIS43LS | Efficacy Study: Arm 1: 10 mg/kg of CIS43LS | Efficacy Study: Arm 2: 40 mg/kg of CIS43LS
Number analyzed (Participants) | 6 | 6 | 6 | 110 | 109
µg/mL | 120.98 (22.41) | 280.52 (40.56) | 897.21 (105.41) | 239.62 (62.77) | 1033.63 (286.52)

8. Secondary Outcome: Time to Maximum Serum Concentration (Tmax) for CIS43LS
Description: Time to maximum total serum concentration (Cmax) of CIS43LS by dose group following a single intravenous administration. Tmax is the time it takes to reach Cmax of CIS43LS after it has been administered; it is determined based on the summary PK curve for each dose group. This was calculated by subtracting the time the CIS43LS intravenous infusion was stopped from the time the blood was collected for the Cmax, at the post-one hour blood draw.
Time Frame: One to 24 hours post-infusion
Population: All participants who received CIS43LS, excluding placebo group.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Dose-escalation Study: Arm 1: 5 mg/kg of CIS43LS | Dose-escalation Study: Arm 2: 10 mg/kg of CIS43LS | Dose-escalation Study: Arm 3: 40 mg/kg of CIS43LS | Efficacy Study: Arm 1: 10 mg/kg of CIS43LS | Efficacy Study: Arm 2: 40 mg/kg of CIS43LS
Number analyzed (Participants) | 6 | 6 | 6 | 110 | 109
Hours | 0.561 (0.040) | 0.556 (0.054) | 0.583 (0.033) | 1.954 (5.390) | 0.597 (0.115)

ADVERSE EVENTS:
Time Frame: Up to 24 weeks
Arm/Group | Dose-escalation Study: Arm 1: 5 mg/kg of CIS43LS | Dose-escalation Study: Arm 2: 10 mg/kg of CIS43LS | Dose-escalation Study: Arm 3: 40 mg/kg of CIS43LS | Efficacy Study: Arm 1: 10 mg/kg of CIS43LS | Efficacy Study: Arm 2: 40 mg/kg of CIS43LS | Efficacy Study: Arm 3: Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 1/110 | 0/110 | 0/110
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 1/110 | 1/110 | 2/110
Other Adverse Events (participants affected / at risk) | 4/6 | 5/6 | 4/6 | 49/110 | 40/110 | 61/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose-escalation Study: Arm 1: 5 mg/kg of CIS43LS (N=6) | Dose-escalation Study: Arm 2: 10 mg/kg of CIS43LS (N=6) | Dose-escalation Study: Arm 3: 40 mg/kg of CIS43LS (N=6) | Efficacy Study: Arm 1: 10 mg/kg of CIS43LS (N=110) | Efficacy Study: Arm 2: 40 mg/kg of CIS43LS (N=110) | Efficacy Study: Arm 3: Placebo (N=110)
Appendectomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1
Inguinal Hernia Repair (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0
Umbilical Hernia Repair (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1
Hypersplenism (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose-escalation Study: Arm 1: 5 mg/kg of CIS43LS (N=6) | Dose-escalation Study: Arm 2: 10 mg/kg of CIS43LS (N=6) | Dose-escalation Study: Arm 3: 40 mg/kg of CIS43LS (N=6) | Efficacy Study: Arm 1: 10 mg/kg of CIS43LS (N=110) | Efficacy Study: Arm 2: 40 mg/kg of CIS43LS (N=110) | Efficacy Study: Arm 3: Placebo (N=110)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 7 | 2 | 2
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 10 | 17 | 12
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 12 | 12 | 19
Eye Swelling (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Visual Acuity Reduced (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 2 | 3
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 1 | 0 | 4 | 5 | 4
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dental Caries (Gastrointestinal disorders) | 2 | 0 | 1 | 11 | 8 | 4
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0 | 2 | 4 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Food Poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastric Disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Gastric Ulcer (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 2 | 1 | 0 | 14 | 10 | 20
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Gingival Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gingival Ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Mouth Ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 3 | 2 | 2
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Strangulated Umbilical Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 5 | 1 | 4
Umbilical Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2 | 1
Asthenia (General disorders) | 1 | 1 | 2 | 2 | 2 | 1
Chest Discomfort (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chest Pain (General disorders) | 0 | 0 | 1 | 0 | 1 | 4
Chills (General disorders) | 0 | 0 | 1 | 8 | 9 | 12
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hernia Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 2 | 4 | 8 | 11
Swelling (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Acarodermatitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 2 | 1 | 0 | 4 | 2
Dysentery (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Furuncle (Infections and infestations) | 0 | 0 | 0 | 2 | 3 | 5
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Genital Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 5 | 3
Genitourinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Herpes Dermatitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Localised Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Malaria (Infections and infestations) | 3 | 2 | 2 | 26 | 16 | 61
Paronychia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 2
Rhinitis (Infections and infestations) | 4 | 5 | 4 | 18 | 18 | 18
Salmonellosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Sinobronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 1
Tinea Pedis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Tinea Versicolour (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1
Typhus (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 1 | 1 | 2 | 0 | 1
Wound Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0
Limb Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 1
Skin Abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2 | 2 | 2
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 1
Blood Creatinine Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood Pressure Diastolic Decreased (Investigations) | 0 | 0 | 1 | 0 | 1 | 2
Blood Pressure Diastolic Increased (Investigations) | 1 | 1 | 0 | 8 | 4 | 12
Blood Pressure Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood Pressure Systolic Decreased (Investigations) | 0 | 0 | 0 | 2 | 3 | 1
Blood Pressure Systolic Increased (Investigations) | 0 | 0 | 0 | 2 | 5 | 8
Platelet Count Decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 1
White Blood Cell Count Decreased (Investigations) | 0 | 0 | 0 | 7 | 10 | 8
White Blood Cell Count Increased (Investigations) | 0 | 0 | 0 | 0 | 3 | 3
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 3 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 5 | 7 | 5
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4 | 9 | 6
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 | 4 | 10 | 8
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 7 | 4 | 8
Head Discomfort (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 3 | 5 | 4 | 45 | 40 | 51
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 2 | 4 | 1
Breast Pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 2 | 0 | 2
Vaginal Discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 9 | 11 | 14
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 3 | 2
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 3 | 49 | 25 | 32
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 4 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tooth Extraction (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0
Venipuncture (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 2 | 2
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-13): https://cdn.clinicaltrials.gov/large-docs/04/NCT04329104/Prot_SAP_000.pdf